CLINICAL TRIAL: NCT06924749
Title: Study of of Oxygen Nebulized Inhalation EGCG in Cancer Patients With New Coronary：Phase II Clinical Trial
Brief Title: Study of of Oxygen Nebulized Inhalation EGCG in Cancer Patients With New Coronary Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Principal investigator, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTEEC2023
Record Dates: First submitted 2023-08-22; First posted 2025-04-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia, Interstitial; Cancer Patients
Keywords: EGCG
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: CT evaluations were performed by a separate radiologist blinded to both treatment allocation and potential imaging artifacts. Subjective endpoints (e.g., COVID-19 symptoms) were collected via patient self-reporting, entirely recorded by the participants themselves to minimize human interference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGCG#Epigallocatechin-3-gallate # (Experimental): Patients randomized to the EGCG group received nebulized EGCG (5878 µmol/L, 10 mL three times daily) plus standard care. The EGCG formulation (HPLC purity ≥98%, Ningbo Hepu Biotechnology Co., Ltd.) was prepared as a 0.9% normal saline solution for nebulization. The protocol-defined treatment duration was 7 days, with optional patient-directed continuation for up to 14 days or until initiation of anti-tumor therapy, whichever occurred first.
  Interventions: Drug: EGCG
- Conventional Treatment Group (No Intervention): The Conventional Treatment Group was treated with the existing standard drugs.

INTERVENTIONS:
Drug: EGCG — EGCG (high pressure liquid chromatographic purity
  ≥ 95%; from Ningbo Hepu Biotechnology Co., Ltd.) is dissolved in 0.9% normal saline; 10ml is inhaled by atomization three times a day.
  Other Names: epigallocchin-3-gallate
  Arms: EGCG#Epigallocatechin-3-gallate #

SUMMARY:
Epigallocatechin-3-gallate (EGCG) is a major polyphenol of green tea that possesses a wide variety of actions, such as anti-inflammatory, anti-fibrotic, pro-apoptotic, anti-tumorous, and metabolic effects via modulation of a variety of intracellular signaling cascades. In addition, preclinical studies have also emphasized the antiviral activity of epigallocatechin-3-gallate (EGCG), including SARS-CoV-2. In previous studies, we found that EGCG can prevent and cure radiation- induced normal tissue damage in tumor patients. In clinical studies, we found that EGCG can prevent and treat radiation-induced acute radiation esophagitis, acute radiation skin injury, acute radiation oral mucositis with high safety. At the same time, the phase I clinical trial designed by us has confirmed the safety and efficacy of EGCG in the treatment of interstitial pneumonia.

DETAILED DESCRIPTION:
The Phase II study was conducted with a randomized, controlled, placebo dose determined by Phase I. the subjects were divided into two groups (experimental group and placebo group). To observe the effectiveness of EGCG, the researchers will use both clinician assessment and patient self-assessment. Primary endpoint: change in imaging (chest CT) before and after treatment. Secondary evaluation endpoints: 1 Further evaluation of the safety of EGCG. 2 The degree of symptom improvement . 3 Changes in laboratory testing indicators.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed malignant tumors by pathology or cytology
* COVID-19 with a confirmed positive polymerase chain reaction or antigen test result for SARS-CoV-23
* moderate-to-severe COVID-19 pneumonia (defined as any radiographic evidence of pulmonary infiltrates and oxygen saturation >94% on room air)
* Pulmonary function of the patient can be treated with aerosol inhalation for 7 days

Exclusion Criteria:

* Current or recent progresses rapidly and may develop into a Critical illness with coronavirus in a short period of time
* Caused by other viruses such as cytomegalovirus, as well as pneumocystis pneumonia, pulmonary edema, aspiration pneumonia and acute interstitial pneumonia
* Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator would preclude the participant from adhering to the protocol or would increase the risk associated with study participation
* known allergy or hypersensitivity to EGCG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
CT imaging improvement rate of COVID-19 | Baseline before treatment and 7±3 days after treatment
  The number of patients with various outcomes in the two groups was assessed. CT scans were performed before and after treatment, and evaluations of improvement, stability, and deterioration were made according to the assessment criteria from previous studies.

SECONDARY OUTCOMES:
Safety evaluations | baseline and up to 7 days post-treatment
  The incidence of adverse events between the two groups was evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Symptom resolution of COVID-19 | baseline and up to 7 days post-treatment
  Differences in COVID-19 Symptom Scores Between the Two Groups Patients assessed the severity of COVID-19-related symptoms daily using a 4-point scale (0: no symptoms, 1: mild symptoms, 2: moderate symptoms, 3: severe symptoms).
Symptom resolution of COVID-19 | Baseline before treatment and 7 days after treatment
  The number of patients with various COVID-19 symptom outcomes in the two groups was assessed. At the final evaluation, patients compared their symptoms with the baseline to determine whether the symptoms had remained stable, improved, or worsened.

OTHER OUTCOMES:
Changes in hematological biomarkers | Baseline before treatment and 7±3 days after treatment
  Hematological biomarkers such as lactate dehydrogenase, lymphocyte count, platelet count, D-dimer, C-reactive protein, aspartate aminotransferase, alanine aminotransferase, creatinine, procalcitonin , and creatine kinase have previously been identified as associated with clinical outcomes in COVID-19. The levels of these biomarkers were tested using biochemical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Ligang, MD,PhD, Study Chair — Shandong Cancer Hospital and Institute
Locations (2):
- China (2):
  - Shan Dong cancer hospital and institute, Jinan, Shandong
  - Hanxi Zhao, Jinan, Shandong